CLINICAL TRIAL: NCT06533527
Title: Randomized Trial of Holding vs. Continuing Incretin-based Therapies Before Upper Endoscopy
Brief Title: Holding vs. Continuing Incretin-based Therapies Before Upper Endoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Shah,Tilak, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 24-301
Record Dates: First submitted 2024-06-27; First posted 2024-08-01 (Actual); Results first posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus, Type 2; Obesity; Gastroparesis
Keywords: incretin; wegovy; ozempic; mounjaro; glp1; gastroparesis; residual gastric volume; endoscopy; anesthesia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Gastroparesis | interventions — Tirzepatide; semaglutide; Liraglutide; dulaglutide

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Continue medication as normal prior to endoscopic procedure (Active Comparator): Does not withhold incretin therapy, maintains dose/frequency/duration of medication.
  Interventions: Drug: GLP-1 medication
- Hold dose prior to endoscopic procedure (No Intervention): Withholds prior dose of incretin therapy per ASA guidance recommendations.

INTERVENTIONS:
Drug: GLP-1 medication — Continue taking GLP-1 as normally scheduled prior to endoscopy.
  Other Names: Tirzepatide; Semaglutide; Liraglutide; Dulaglutide
  Arms: Continue medication as normal prior to endoscopic procedure

SUMMARY:
To assess whether holding incretin-based therapy before endoscopy reduces the likelihood of clinically relevant Residual Gastric Volume (RGV).

Primary Outcomes:

* Residual gastric volume that precludes adequate endoscopic examination
* Residual gastric volume that necessitates premature termination of the endoscopy procedure
* Need for endotracheal intubation due to stomach contents.
* Occurrence of aspiration events requiring extended observation/monitoring, unplanned therapeutics, and/or hospital admission

Secondary Outcomes:

* Presence of any solid food
* Presence of moderate liquid content
* Increased RGV(Residual Gastric Volume) defined as any amount of solid content or > 0.8 mL/Kg of fluid content (measured from the aspiration/suction canister).
* Differences in primary and secondary outcomes between different medications

ELIGIBILITY:
Inclusion Criteria:

* Patients using incretin-based therapies at a stable dose for more than 1 month.
* Patients scheduled for outpatient esophagogastroduodenoscopy (EGD), endoscopic ultrasound (EUS), or endoscopic retrograde cholangiopancreatography (ERCP) under monitored anesthesia care.

Exclusion Criteria:

* Documented history of gastroparesis (based on a 4-hour solid-phase gastric emptying study)
* Known history of achalasia
* Surgical or genetically altered foregut anatomy
* Known gastric outlet obstruction or pre-procedure imaging suggestive of gastric outlet obstruction.
* Patients who did not follow the standard NPO (nil per oral) instructions.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2024-07-31 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Cleveland Clinic, Weston, Florida
  - Cleveland Clinic, Cleveland, Ohio

REFERENCES:
- [Result] Kobori T, Onishi Y, Yoshida Y, Tahara T, Kikuchi T, Kubota T, Iwamoto M, Sawada T, Kobayashi R, Fujiwara H, Kasuga M. Association of glucagon-like peptide-1 receptor agonist treatment with gastric residue in an esophagogastroduodenoscopy. J Diabetes Investig. 2023 Jun;14(6):767-773. doi: 10.1111/jdi.14005. Epub 2023 Mar 15. PMID 36919944
- [Result] Silveira SQ, da Silva LM, de Campos Vieira Abib A, de Moura DTH, de Moura EGH, Santos LB, Ho AM, Nersessian RSF, Lima FLM, Silva MV, Mizubuti GB. Relationship between perioperative semaglutide use and residual gastric content: A retrospective analysis of patients undergoing elective upper endoscopy. J Clin Anesth. 2023 Aug;87:111091. doi: 10.1016/j.jclinane.2023.111091. Epub 2023 Mar 2. PMID 36870274
- [Result] Joshi G, Abdelmalak B, Weigel W, et al. American Society of Anesthesiologists Consensus-Based Guidance on Preoperative Management of Patients (Adults and Children) on Glucagon-Like Peptide-1 (GLP-1) Receptor Agonists. Released June 29, 2023. Accessed from asahq.org on January 16, 2024.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adults 18 or older who were scheduled to undergo an upper endoscopic procedure under monitored anesthesia care or moderate sedation were recruited from Cleveland Clinic hospital main campus or Cleveland Clinic Weston. Patients undergoing colonoscopy were permitted to participate if they were also undergoing an upper endoscopic procedure concurrently. Recruitment occurred from July 2024 until May 2025.
Pre-assignment Details: One patient was excluded prior to assignment due to having stop the GLP medication prior to randomization.
Period: Overall Study
Arm/Group | Continue medication as normal prior to endoscopic procedure | Hold dose prior to endoscopic procedure
Started | 28 | 32
Completed | 28 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Nine patients met exclusion criteria and not included in analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Continue Medication as Normal Prior to Endoscopic Procedure | Hold Dose Prior to Endoscopic Procedure | Total
Number analyzed (Participants) | 28 | 32 | 60
Age, Continuous [Median (Full Range); unit: years] | 62.5 [30 to 87] | 62.5 [39 to 78] | 62.5 [30 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 13 | 17 | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Diabetes [Count of Participants; unit: Participants] — Population: Number of patients with diagnosed with Diabetes Mellitus
  Participants | 7 | 10 | 17
A1c greater than 7 [Count of Participants; unit: Participants] — Percent of glycated hemoglobin
  Participants | 7 | 6 | 13
A1c [Median (Full Range); unit: Percent of glycated hemoglobin] — Median A1c of participants
  Percent of glycated hemoglobin | 6.4 [5 to 10.6] | 6.4 [4.8 to 9.2] | 6.4 [4.8 to 10.6]
BMI [Median (Full Range); unit: kg/m^2] | 31.0 [20.2 to 40.9] | 29.7 [23.6 to 49.9] | 30 [20.2 to 49.9]
Drug type [Count of Participants; unit: Participants] — What GLP medication is patient taking
  Participants
    Dulaglutide | 3 | 4 | 7
    Semaglutide | 10 | 20 | 30
    Tirzepatide | 15 | 8 | 23
Duration on drug [Median (Full Range); unit: months] — Length of time patient has been taking GLP-1 medication (months)
  months | 6.0 [1 to 70] | 5.5 [1 to 48] | 5.8 [1 to 70]
Indications for the Procedure [Count of Participants; unit: Participants] — Some participants may have multiple indications for the procedure while some may have no indication. This results in a difference between the total number of participants and the number of indications reported.
  Participants
    Heartburn | 3 | 5 | 8
    Dyspepsia | 3 | 2 | 5
    Anemia | 1 | 0 | 1
    Disease follow-up | 8 | 12 | 20
    Others | 10 | 13 | 23
Preprocedural symptoms [Count of Participants; unit: Participants]
  Nausea | 1 | 0 | 1
  Vomiting | 1 | 0 | 1
  Heartburn | 1 | 0 | 1
  Dyspepsia | 1 | 1 | 2
  Bloating | 2 | 1 | 3
  Other Symptoms | 9 | 12 | 21
  No symptoms reported | 13 | 18 | 31

OUTCOME MEASURES:

1. Primary Outcome: Presence of RGV (Residual Gastric Volume) in Stomach
Description: Residual gastric volume (RGV) that precludes adequate endoscopic examination
Time Frame: Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Continue medication as normal prior to endoscopic procedure | Hold dose prior to endoscopic procedure
Number analyzed (Participants) | 28 | 32
Participants | 7 | 1

2. Primary Outcome: Tracking the Use of Intubation Due to RGV
Time Frame: Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Continue medication as normal prior to endoscopic procedure | Hold dose prior to endoscopic procedure
Number analyzed (Participants) | 28 | 32
Participants | 0 | 0

3. Primary Outcome: Aspiration Events Due to RGV (Residual Gastric Volume)
Description: Occurrence of aspiration events requiring extended observation/monitoring, unplanned therapeutics, and/or hospital admission
Time Frame: Procedure
Measure: Number; unit: number of aspiration events
Arm/Group | Continue medication as normal prior to endoscopic procedure | Hold dose prior to endoscopic procedure
Number analyzed (Participants) | 28 | 32
number of aspiration events | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events collected from the time of the endoscopy procedure up to one week after the procedure.
Arm/Group | Continue medication as normal prior to endoscopic procedure | Hold dose prior to endoscopic procedure
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/32
Other Adverse Events (participants affected / at risk) | 0/28 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan: Protocol Ver. 5 (2025-02-03): https://cdn.clinicaltrials.gov/large-docs/27/NCT06533527/Prot_SAP_001.pdf